CLINICAL TRIAL: NCT01794052
Title: m-Power Heart Project
Brief Title: To Develop a High Quality Health Care Delivery Model for the Management of Hypertension and Diabetes at CHCs and District Hospitals of Himachal Pradesh.
Acronym: m-Power Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Chronic Disease Control, India (Other)
Collaborators: All India Institute of Medical Sciences (Other); Public Health Foundation of India (Other)
Responsible Party: Principal Investigator, Dr. Dorairaj Prabhakaran, Executive Director, Centre for Chronic Disease Control, India
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CCDC-2013/001; CTRI/2013/02/003412 (Registry Identifier: Clinical Trials Registry India)
Record Dates: First submitted 2013-01-23; First posted 2013-02-18 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-08

CONDITIONS: Hypertension; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DSS enabled health care delivery model (Experimental): Evidence based, DSS enabled, health care delivery model
  Interventions: Other: Evidence based, DSS enabled, health care delivery model

INTERVENTIONS:
Other: Evidence based, DSS enabled, health care delivery model — The study focus on preliminary work before a definitive randomised controlled trial. In this phase, we are developing an intervention for the evidence based management of hypertension and diabetes at primary care setting in India.
  The components of the interventions that we are developing are:
  1. A structured training of the health care staff for identifying people at risk of developing diabetes or hypertension
  2. Treating patients as per a standard clinical guidelines
  3. Giving health education to patients on lifestyle changes for better self-care
  4. Optimizing the care pathways at the health facilities to enable better delivery of the intervention and
  5. Development and implementation of a smartphone based decision support system (DSS) with inbuilt diagnostic and treatment algorithm

SUMMARY:
Hypertension and diabetes are major risk factors for cardiovascular diseases. Although these two conditions can be detected much early in life and are amenable to interventions at primary health care level, the health system in India fails to provide adequate interventions at primary health care level which translates to huge burden of undiagnosed and uncontrolled hypertension and diabetes in the community. This study aims to design a feasible and sustainable evidence-based, decision support-enabled, health care delivery model for the management of hypertension and diabetes in the primary health care facilities of Himachal Pradesh. The study will be conducted at the 5 Community Health Centers (CHCs) and District Hospital of Solan District, Himachal Pradesh using both qualitative and quantitative methods. The design and development of the model will be carried out in the initial six months followed by piloting the services at the CHCs and District Hospital. The impact of the model on quality of care will be assessed in a pre-post design measuring changes in both clinical and process indicators.

DETAILED DESCRIPTION:
This study aims to design a feasible and sustainable evidence-based, decision support-enabled, health care delivery model for the management of hypertension and diabetes in the primary health care facilities of Himachal Pradesh. The study will be conducted at the 5 Community Health Centers (CHCs) and District Hospital of Solan District, Himachal Pradesh using both qualitative and quantitative methods. The design and development of the model will be carried out in the initial six months followed by piloting the services at the CHCs and District Hospital. The impact of the model on quality of care will be assessed in a pre-post design measuring changes in both clinical and process indicators.

ELIGIBILITY:
Inclusion Criteria:

* All consenting adults of age >30 years attending the Community Health Centre's and Civil Hospital of Solan District of Himachal Pradesh.

Exclusion Criteria:

* Person not willing to consent
* <30 years of age
* History of coronary heart disease or stroke
* Pregnant OR trying to become pregnant OR of child-bearing potential and not actively practicing birth control (including natural methods)
* Malignancy or life-threatening diseases

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6797 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in the proportion of people with hypertension and/or diabetes receiving evidence based clinical management. | 30 months
Change in compliance to therapy and follow-up rate among people with hypertension and/or diabetes. | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Dorairaj Prabhakaran, MD, DM, MSc, FRCP, Principal Investigator — Centre for Chronic Disease Control
Locations (1):
- CHCs and District Hospital of Solan District, Solan, Himachal Pradesh, India

REFERENCES:
- [Derived] Ajay VS, Jindal D, Roy A, Venugopal V, Sharma R, Pawar A, Kinra S, Tandon N, Prabhakaran D. Development of a Smartphone-Enabled Hypertension and Diabetes Mellitus Management Package to Facilitate Evidence-Based Care Delivery in Primary Healthcare Facilities in India: The mPower Heart Project. J Am Heart Assoc. 2016 Dec 21;5(12):e004343. doi: 10.1161/JAHA.116.004343. PMID 28003248